CLINICAL TRIAL: NCT04993937
Title: Effectiveness of 6 Weeks Plyometric Training on Agility Among University Male Students.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC/00925 Nadeem Asghar
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Sports Physical Therapy
Keywords: T test,; Ilinois agility test,; Plyometric training
MeSH Terms: interventions — Methods; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group will follow their daily routine activities.
  Interventions: Other: Control Group
- Experimental group (Experimental): Interventional group will receive 6 weeks of plyometric training and receive training for week and three sessions in a week.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Interventional group will receive 6 weeks of plyometric training and receive training for week and three sessions in a week.
  Arms: Experimental group
Other: Control Group — Control group will follow their daily routine activities and may involve in any other exercise program rather than plyometric exercises.
  Arms: Control group

SUMMARY:
Plyometrics is a kind of exercise training that focuses on increasing muscular power by varying the pace and force of various motions. Plyometrics training can help you enhance your physical performance and ability to do a variety of tasks. Pushups, throwing, sprinting, leaping, and kicking are just a few examples of plyometric activities. Plyometrics are commonly used by athletes, although these routines may be done by anybody. Plyometrics are used by people in physical therapy after an accident or injury to get back into form and physical function. Speed, explosive power, coordination, and particular sports skills may all be improved with agility training. Agility training routines can benefit players of all levels, from high school to professional sports teams. Include these drills in your training regimen a few times a week to improve your foot speed and sports technique.

DETAILED DESCRIPTION:
The ability of the neuromuscular and musculoskeletal systems to generate force at a specific velocity, in a particular direction, appears to be critical for many sports that involve sprinting, jumping and throwing. In light of the above, plyometric training can be used to enhance the ability of skeletal muscle to exert maximal force in as short a time as possible. Plyometric training typically includes various unilateral and bilateral jumps, hops and bounds with coaches often prescribing these in a multidirectional fashion to reflect the unpredictable nature of field and court sports. The rationale of this approach is founded on the well-accepted principle that adaptations to vertically (VPT) and horizontally orientated PT will transfer better to athletic tasks that are carried out in the same direction as they are performed. Plyometric consists of a rapid stretching of a muscle (eccentric action) immediately followed by a concentric or shortening action of the same muscle and connective tissue, the stored elastic energy within the muscle is used to produce more force than can be provided by a concentric action alone. Though aerobic capacity is important during a soccer game high-intensity single-bout efforts also play an important role for physical performance. in this sense, aside from endurance activity, female soccer players must also perform numerous explosive action including jumping, kicking, accelerating, decelerating and changing of direction, with most of these preceding goal opportunities in competitive leagues. specifically, the straight sprint (45%) followed by vertical jumps (16%) have shown to be the two most frequent actions in goal situations during professional soccer matches. Studies also suggest that changes in motor performance skills resulting from the performance of combined resistance training and plyometric training are greater than with either type of training alone. Six weeks of combined resistance training and plyometric training would lead to greater improvements in fitness performance in healthy boys than resistance training and static stretching. Plyometric training has been proposed for the development of explosive power performance and specifically for the improvement of vertical jump ability. he main finding of this study was the improvement of either vertical- and horizontal jump performance in basketball players as a consequence of a multipurpose plyometric training intervention.

ELIGIBILITY:
Inclusion Criteria:

* Students will be selected that have spent at least one year
* BMI (18.5 to 24.9 kg/m2)
* Only male students will be included

Exclusion Criteria:

* Students undergone surgery or had accident within last 6 months.
* Should not involve in any plyometric technique before and at the time of study
* Students involved in any other exercise plan
* Not willing students

Ages: 19 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
T test | 6th day
  In T test players have to run 40 yards and time will be noted in seconds. Rating starts from >11.5 seconds (poor) to <9.5 seconds (excellent).
Illinois agility test | 6th day
  Player have to run about 60 meters and time will be noted in seconds with rating poor >18.8 seconds and excellent <15.9 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Danish Latif, MSPT-SPT, Principal Investigator — Riphah International University
Locations (1):
- University of Lahore, Chenab Campus, Gujrat, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Izquierdo M, Hakkinen K, Gonzalez-Badillo JJ, Ibanez J, Gorostiaga EM. Effects of long-term training specificity on maximal strength and power of the upper and lower extremities in athletes from different sports. Eur J Appl Physiol. 2002 Jul;87(3):264-71. doi: 10.1007/s00421-002-0628-y. Epub 2002 May 22. PMID 12111288
- [Background] Loturco I, Pereira LA, Kobal R, Zanetti V, Kitamura K, Abad CC, Nakamura FY. Transference effect of vertical and horizontal plyometrics on sprint performance of high-level U-20 soccer players. J Sports Sci. 2015;33(20):2182-91. doi: 10.1080/02640414.2015.1081394. Epub 2015 Sep 21. PMID 26390150
- [Background] Chmielewski TL, Myer GD, Kauffman D, Tillman SM. Plyometric exercise in the rehabilitation of athletes: physiological responses and clinical application. J Orthop Sports Phys Ther. 2006 May;36(5):308-19. doi: 10.2519/jospt.2006.2013. PMID 16715831
- [Background] Ramirez-Campillo R, Alvarez C, Garcia-Hermoso A, Ramirez-Velez R, Gentil P, Asadi A, Chaabene H, Moran J, Meylan C, Garcia-de-Alcaraz A, Sanchez-Sanchez J, Nakamura FY, Granacher U, Kraemer W, Izquierdo M. Methodological Characteristics and Future Directions for Plyometric Jump Training Research: A Scoping Review. Sports Med. 2018 May;48(5):1059-1081. doi: 10.1007/s40279-018-0870-z. PMID 29470823
- [Background] Ziv G, Lidor R. Vertical jump in female and male basketball players--a review of observational and experimental studies. J Sci Med Sport. 2010 May;13(3):332-9. doi: 10.1016/j.jsams.2009.02.009. Epub 2009 May 13. PMID 19443269
- [Background] Ziv G, Lidor R. Vertical jump in female and male volleyball players: a review of observational and experimental studies. Scand J Med Sci Sports. 2010 Aug;20(4):556-67. doi: 10.1111/j.1600-0838.2009.01083.x. PMID 20459471
- [Background] Cappa DF, Behm DG. Training specificity of hurdle vs. countermovement jump training. J Strength Cond Res. 2011 Oct;25(10):2715-20. doi: 10.1519/JSC.0b013e318208d43c. PMID 21873903
- [Background] Miller MG, Herniman JJ, Ricard MD, Cheatham CC, Michael TJ. The effects of a 6-week plyometric training program on agility. J Sports Sci Med. 2006 Sep 1;5(3):459-65. eCollection 2006. PMID 24353464
- [Background] Thomas K, French D, Hayes PR. The effect of two plyometric training techniques on muscular power and agility in youth soccer players. J Strength Cond Res. 2009 Jan;23(1):332-5. doi: 10.1519/JSC.0b013e318183a01a. PMID 19002073
- [Background] Vaczi M, Tollar J, Meszler B, Juhasz I, Karsai I. Short-term high intensity plyometric training program improves strength, power and agility in male soccer players. J Hum Kinet. 2013 Mar 28;36:17-26. doi: 10.2478/hukin-2013-0002. Print 2013 Mar. PMID 23717351
- [Background] Faigenbaum AD, McFarland JE, Keiper FB, Tevlin W, Ratamess NA, Kang J, Hoffman JR. Effects of a short-term plyometric and resistance training program on fitness performance in boys age 12 to 15 years. J Sports Sci Med. 2007 Dec 1;6(4):519-25. eCollection 2007. PMID 24149486
- [Background] Khlifa R, Aouadi R, Hermassi S, Chelly MS, Jlid MC, Hbacha H, Castagna C. Effects of a plyometric training program with and without added load on jumping ability in basketball players. J Strength Cond Res. 2010 Nov;24(11):2955-61. doi: 10.1519/JSC.0b013e3181e37fbe. PMID 20938357
- [Background] Foure A, Nordez A, Cornu C. Plyometric training effects on Achilles tendon stiffness and dissipative properties. J Appl Physiol (1985). 2010 Sep;109(3):849-54. doi: 10.1152/japplphysiol.01150.2009. Epub 2010 Jun 24. PMID 20576842
- [Background] Ramirez-Campillo R, Andrade DC, Izquierdo M. Effects of plyometric training volume and training surface on explosive strength. J Strength Cond Res. 2013 Oct;27(10):2714-22. doi: 10.1519/JSC.0b013e318280c9e9. PMID 23254550
- [Background] di Cagno A, Iuliano E, Buonsenso A, Giombini A, Di Martino G, Parisi A, Calcagno G, Fiorilli G. Effects of Accentuated Eccentric Training vs Plyometric Training on Performance of Young Elite Fencers. J Sports Sci Med. 2020 Nov 19;19(4):703-713. eCollection 2020 Dec. PMID 33239944
- [Background] Diallo O, Dore E, Duche P, Van Praagh E. Effects of plyometric training followed by a reduced training programme on physical performance in prepubescent soccer players. J Sports Med Phys Fitness. 2001 Sep;41(3):342-8. PMID 11533565